CLINICAL TRIAL: NCT03379714
Title: Data Collection of the Treatment of Intracranial Aneurysms With the WEB™ Aneurysm Embolization System: a Monocentric Post-market Observational Study
Brief Title: Mid-term Data Collection of the Treatment of Intracranial Aneurysms With the WEB™ Aneurysm Embolization System
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision
Sponsor: Medical Therapy Solutions (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Other Study IDs: MTS-02
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2017-12

CONDITIONS: Ruptured and Unruptured Intracranial Aneurysms
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ruptured or unruptured intracranial aneurysms
  Interventions: Device: WEB aneurysm embolization system

INTERVENTIONS:
Device: WEB aneurysm embolization system — The WEB aneurysm embolization system is a class III device and consists of an implantable embolization device attached to a delivery device. The WEB is a mesh composed of single layers of braided nitinol tubes with platinum cores. The braids are held together by proximal and distal platinum/ iridium radiopaque markers.

SUMMARY:
Flow disruption is a new endovascular approach for treatment of both ruptured and unruptured intracranial aneurysms, which involves placement of an endosaccular device (WEB) which modifies the blood flow at the level of the neck and induces intraaneurysmal thrombosis. The WEB was designed to treat wide-neck bifurcation aneurysms. This observational study will collect data about the routine practice in one center of using the WEB in ruptured and unruptured intracranial aneurysms. The primary objective is to evaluate its efficacy by assessing the anatomic outcome during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. Patient is capable to undergo general anaesthesia.
3. Patient must sign and date the informed consent form prior to data registration. If patient is not able to give informed consent for himself/herself, a legally authorized representative must give informed consent on his/her behalf.
4. Patient has a ruptured or unruptured intracranial aneurysm requiring endovascular treatment.
5. Aneurysm with dome-to-neck ratio ≥ 1.
6. Aneurysm size favourable for WEB implantation (aneurysm width < 10 mm or aneurysm width > 3mm).

Exclusion Criteria:

1. Patient is pregnant.
2. Patient has renal insufficiency (GRF < 45 ml/min/1.73 m2).
3. Patient is unable to comply with the study protocol (e.g. no permanent address, known to be non-compliant or presenting an unstable psychiatric history).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ruptured or unruptured intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of anatomic outcome | at 6 months
  grade of occlusion of the aneurysm assessed by MRA
  WEB Occlusion Scale:
  WOS A: complete occlusion WOS B: complete occlusion with opacification of the proximal recess WOS C: residual neck filling WOS D: residual aneurysm filling
Determination of anatomic outcome | at 24 months
  grade of occlusion of the aneurysm assessed by MRA
  WEB Occlusion Scale:
  WOS A: complete occlusion WOS B: complete occlusion with opacification of the proximal recess WOS C: residual neck filling WOS D: residual aneurysm filling

SECONDARY OUTCOMES:
Determination of procedural complications (Adverse events) during the operation | during index-procedure
  Procedural complications: aneurysm rupture, dissection, thromboembolic events (symptomatic and non-symptomatic), device protrusion through the neck of the aneurysm inside the parent artery, detachment problem, device stuck in microcatheter, bleeding.
Recording the use of additional devices during treatment. | during index-procedure
  Possible additional devices are stent, coils, flow diverter
Determination of the occurrence of post-procedural symptomatic thromboembolic events | up to 24 months follow-up
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | At baseline
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 6 to 8 weeks follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 6 months follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Determination of clinical outcome: assessing disability of the patient by the modified Rankin Scale (mRS) | at 24 months follow-up
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Fisher grade (severity of intracranial SAH) for ruptured aneurysms. | at baseline
  Fisher grade:
  1 No haemorrhage evident. 2 Subarachnoid haemorrhage less than 1mm thick. 3 Subarachnoid haemorrhage more than 1mm thick. 4 Subarachnoid haemorrhage of any thickness with intraventricular haemorrhage (IVH) or parenchymal extension.
Determination of technical success of the device | during index-procedure
  Technical success is defined as device deployment in the target aneurysm as intended by the investigator with adequate occlusion of the aneurysm (WOS A, B or C).
Determination of overall mortality | up to 24 months
Recording of intracranial haemorrhage during follow-up | up to 24 months
Recording the need for re-intervention during follow-up. | up to 24 months
Hunt and Hess scale (severity of clinical effect of SAH) for ruptured aneurysms. | baseline
  Hunt and Hess scale:
  1. asymptomatic or minimal headache and slight neck stiffness, 70% survival
  2. moderate to severe headache; neck stiffness; no neurologic deficit except cranial nerve palsy; 60% survival
  3. drowsy; minimal neurologic deficit; 50% survival
  4. stuporous; moderate to severe hemiparesis; possibly early decerebrate rigidity and vegetative disturbances; 20% survival
  5. deep coma; decerebrate rigidity; moribund;10% survival

CONTACTS AND LOCATIONS:
Overall Officials: Maurits Voormolen, Prof Dr, Principal Investigator — Study Principal Investigator
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No